CLINICAL TRIAL: NCT00262626
Title: A Multicentre Study on the Risk Factors for the Progression of Open-Angle Glaucoma
Brief Title: The Canadian Glaucoma Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Dalhousie University (Other)
Collaborators: Canadian National Institute for the Blind (Other); Glaucoma Research Society of Canada (Other); Allergan (Industry); Merck Frosst Canada Ltd. (Industry); Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CGS1
Record Dates: First submitted 2005-12-05; First posted 2005-12-07 (Estimated); Last update posted 2005-12-07 (Estimated); Status verified 2003-06

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma | interventions — Trabeculectomy

INTERVENTIONS:
Drug: Intraocular pressure reduction
Procedure: Argon laser trabeculoplasty
Procedure: Trabeculectomy

SUMMARY:
Glaucoma is a disease which affects between one and two percent of all individuals aged over 40 years. According to recent Canadian National Institute for the Blind figures, it is the second largest specific cause of blindness in this country. The most common form of glaucoma, open-angle glaucoma, is incipient and typically results in a progressive loss of vision without symptoms due to damage to a structure inside the eye called the optic nerve head. Although the most important known risk factor for the development of open-angle glaucoma is high intraocular pressure (the pressure within the eyeball), a number of researchers have shown that a sizeable proportion of patients continue to lose vision in spite of successful treatment to lower their intraocular pressure. This finding suggests that there may be additional risk factors involved. Ocular vasospasm (the inability of certain blood vessels to dilate and increase blood flow according to the needs the eye) and vascular disease are among other factors implicated but their roles have not yet been fully investigated. The Canadian Glaucoma Study Group proposes to investigate the role of risk factors, including vasospasm and vascular disease, involved in the progression of open-angle glaucoma. We will recruit 410 patients with open-angle glaucoma across 4 centres (Halifax, Vancouver, Montreal and Toronto) who will be treated by experienced investigative ophthalmologists according to a uniform standard protocol to ensure that all patients are managed in the same manner. The patients will be followed meticulously with the most modern and accurate tests available every four months for a period of 5 years to determine whether progression has taken place. Visual function will be measured using two techniques called conventional perimetry and blue-on-yellow perimetry, and optic nerve heads will be examined with a special scanner capable of three-dimensional imaging. By defining both the ocular and systemic profiles of patients who progress and do not progress, we may be able to identify which patients will benefit from the standard treatment of intraocular pressure reduction, such as that prescribed in the study. More importantly, we will identify the characteristics of patients who do not benefit from standard treatment, so that alternative ones may be developed. Such studies are clearly necessary, but have not yet been conducted. We believe that the proposed study will increase our knowledge of open-angle glaucoma and reduce its impact on blindness and visual disability.

DETAILED DESCRIPTION:
Elevated intraocular pressure is the most important known risk factor for the development and progression of open-angle glaucoma. While pressure reduction is beneficial in many cases, a significant proportion of patients continue to progress despite clinically acceptable pressure levels. Many investigators have found no differences in pressure characteristics between progressing and non-progressing patients, highlighting our current inability to identify which patients will respond to pressure reduction. It is likely that this inability stems from our poor understanding of the risk factors, both ocular and systemic, for progression and the probability that glaucoma is a disease with multiple pathogenic mechanisms.

In this application the Canadian Glaucoma Study Group proposes a multi-centre prospective study with the objective of characterising the risk factors associated with the progression of open-angle glaucoma. We will determine sub-groups of patients with regard to the type of progression, thereby allowing us to identify the ocular and systemic profiles of patients who are likely to and not likely to benefit from intraocular pressure reduction.

Our hypotheses are:

(i) The relationship between intraocular pressure characteristics during follow-up and survival rates with regard to progression of open-angle glaucoma is weak.

(ii) Patients with vasospasm have a higher survival rate than patients without vasospasm with the clinical management prescribed in this study.

(iii) Patients with vascular disease have a lower survival rate than patients without vascular disease with the clinical management prescribed in this study.

We will test these hypotheses by following a total of 410 patients in 4 centres (Halifax, Vancouver, Montreal and Toronto) every 4 months for a period of 5 years using a uniform protocol for both the clinical management and study procedures. Clinical management will involve at least 30% reduction in intraocular pressure from the baseline untreated value, followed by an additional 20% or greater reduction after a progressive event. The study procedures include conventional perimetry, blue-on-yellow perimetry and scanning laser tomography of the optic nerve head and nerve fibre layer. We will measure finger blood flow with both heat and cold provocation to assess each patient's susceptibility to vasospasm and also obtain haematological, biochemical and rheological profiles to assess the presence of vascular disease.

Progression of either visual field and optic nerve head damage will be termed a progressive event occurring after a predefined change from baseline. Events will be defined separately for each technique based on percentiles of empirically derived values of test-retest variability, allowing a degree of standardisation between techniques. Comparison of survival times between groups (e.g. vasospastic and non-vasospastic) will be made with Cox's survivorship analysis with a repeated measures model. Where appropriate, group comparisons will be made with the group t-test or Mann-Whitney test.

If we can characterise more fully the risk factors for glaucomatous progression, we may be able to identify the ocular and systemic profiles of patients who will benefit from our current treatment of pressure reduction. More importantly, we can identify the profiles of patients who respond poorly to pressure reduction so that future research efforts can lead to the development and implementation of alternative therapy. We believe that this is a significant study which will result in a better understanding of open-angle glaucoma and help reduce its impact on blindness and visual disability.

ELIGIBILITY:
Inclusion Criteria:

1. Best corrected visual acuity of at least 6/9.
2. Previous visual field examinations showing nerve fibre bundle visual field defects characteristic of open-angle glaucoma and/or previous optic nerve head photographs showing cupping or notching characteristic of open-angle glaucoma.
3. Total visual field damage [in the eligibility visual field (see Section 6.1)] of between 2 and 10 dB using the visual field index Mean Deviation.46
4. Access to patient's previous ocular history and availability of initial untreated intraocular pressure (minimum of three readings).

(d) Normal non-closable angles by gonioscopy. (e) Willingness to participate in the study and to give informed consent.

Exclusion Criteria:

1. Non-glaucomatous ocular disease.
2. Systemic disease known to affect the visual field or ability to participate in the study.
3. Systemic beta-blockers.
4. Chronic ocular medication other than for glaucoma.
5. Previous incisional ocular surgery.

(e) Distance refraction exceeding 6.00 diopters equivalent sphere or 2.50 diopters of astigmatism.

(f) Aphakia or pseudophakia. (g) Contact lens wear.

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 430
Dates: Start 1995-02; Study Completion 1995-06

PRIMARY OUTCOMES:
Visual field progression

SECONDARY OUTCOMES:
Optic disc progression

CONTACTS AND LOCATIONS:
Overall Officials: Balwantray C Chauhan, Ph.D., Principal Investigator — Dalhousie University
Locations (4):
- Canada (4):
  - University of British Columbia, Vancouver, British Columbia
  - Dalhousie University, Halifax, Nova Scotia
  - University of Toronto, Toronto, Ontario
  - University of Montreal, Montreal, Quebec

REFERENCES:
- [Derived] Chauhan BC, Mikelberg FS, Artes PH, Balazsi AG, LeBlanc RP, Lesk MR, Nicolela MT, Trope GE; Canadian Glaucoma Study Group. Canadian Glaucoma Study: 3. Impact of risk factors and intraocular pressure reduction on the rates of visual field change. Arch Ophthalmol. 2010 Oct;128(10):1249-55. doi: 10.1001/archophthalmol.2010.196. Epub 2010 Aug 9. PMID 20696979
- [Derived] Chauhan BC, Mikelberg FS, Balaszi AG, LeBlanc RP, Lesk MR, Trope GE; Canadian Glaucoma Study Group. Canadian Glaucoma Study: 2. risk factors for the progression of open-angle glaucoma. Arch Ophthalmol. 2008 Aug;126(8):1030-6. doi: 10.1001/archopht.126.8.1030. PMID 18695095